CLINICAL TRIAL: NCT04342117
Title: PI3K-Inhibitor Registry Study: Real-World Treatment Utilization and Effectiveness of PI3K-inhibitors in Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma and Follicular Lymphoma
Brief Title: Observational Trial of Real-World Treatment Utilization and Effectiveness of PI3K-inhibitors in CLL/SLL and FL
Acronym: REAL
Status: Terminated | Type: Observational
Why Stopped: Strategy Change
Sponsor: SecuraBio (Industry)
Responsible Party: Sponsor
Other Study IDs: VS-0145-401
Record Dates: First submitted 2020-03-24; First posted 2020-04-10 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Lymphoma, Small Lymphocytic; Lymphoma; Lymphoma, Non-Hodgkin; Chronic Lymphocytic Leukemia; Follicular Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, Follicular | interventions — duvelisib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Duvelisib: Patients who take duvelisib.
  Interventions: Drug: duvelisib
- Other PI3K-inhibitors: Patients who take a PI3K-inhibitor other than duvelisib
  Interventions: Drug: PI3K inhibitor

INTERVENTIONS:
Drug: duvelisib — 25 mg BID, 15 mg BID
  Other Names: Copiktra, VS-0145
  Groups: Duvelisib
Drug: PI3K inhibitor — FDA approved PI3K inhibitors
  Groups: Other PI3K-inhibitors

SUMMARY:
This study will assess whether there are differences in effectiveness and safety outcomes among PI3K-treated patients in a real world registry, compared to patients treated in clinical trials.

DETAILED DESCRIPTION:
Phase IV, multicenter, prospective observational study in a real world (RW) setting, designed to observe the utilization and effectiveness of PI3K-inhibitor treatment, and HRQoL of patients with CLL/SLL/FL outside the context of a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Clinical or pathological diagnosis of CLL/SLL according to the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) diagnosis guideline or pathological diagnosis of FL, for whom the Investigator has decided that PI3K-inhibitor treatment is the appropriate therapy

  * Patients previously treated with PI3K-inhibitors are eligible for this study if they:

    * Are restarting treatment with PI3K-inhibitor at enrollment, or
    * Restarted PI3K-inhibitor treatment within 3 treatment cycles prior to enrollment
  * Patients newly treated with PI3K-inhibitors are eligible for this study if they:

    * Are starting treatment with PI3K-inhibitors at enrollment, or
    * Started on PI3K-inhibitor treatment within 3 treatment cycles prior to enrollment
* ≥18 years of age at time consent is provided to participate in this study
* For patients treated with PI3K-inhibitors prior to enrollment in the study, availability of documentation of previous PI3K-inhibitor treatment, including the start date of previous or current PI3K-inhibitor treatment in patient charts or medical records
* Patient is willing and able to provide a signed and dated Institutional Review Board (IRB)-approved informed consent form (ICF)

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 200 patients with a clinical or pathological diagnosis of CLL/SLL or pathological diagnosis of FL, for whom the Investigator has decided PI3K-inhibitor treatment is the appropriate therapy will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Event-Free Survival (EFS) | 2 years
  Observe the effectiveness of the PI3K-inhibitor administered

SECONDARY OUTCOMES:
Measurement of Quality of Life - EQ-5D | 2 years
  EQ-5D is a widely used health status instrument, which developed by the EuroQol Group in the 1980s. It provides a concise and generic measure to compare and value health status across disease areas. The 5-level EQ-5D-5L was introduced in 2009 to improve the sensitivity of the instrument and reduce the ceiling effect. The EQ-5D-5L consists of the descriptive system measuring 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression and the EQ visual analogue scale (VAS). The patient is asked to indicate his/her health state by choosing one of the 5 levels for each dimension: no problem, slight problems, moderate problems, severe problems and extreme problems. Each dimension has a 1-digit number that expresses the level selected for that dimension. The digit for the 5 dimensions will be combined into a 5-digit number that describes a patient's health profile. Results of the EQ VAS will be presented to measure overall self-rated health status.
Measurement of Quality of Life - FACT-lym | 2 years
  The Functional Assessment of Cancer Therapy - Lymphoma (FACT-lym) is a PRO measure used to assess HRQoL in patients undergoing cancer therapy. The instrument includes 27 questions on the impacts of cancer therapy over the past 7 days in four domains plus 15 questions related to lymphoma patients: physical, social/family, emotional, and functional over the past 7 days. Each question is answered using a 5-point Likert scale ranging from 0 (not at all) to 4 (very much), where higher numbers indicate better health state. Scores of each domain will be calculated by adding scores for questions included in each domain, and a total score for the FACT-Lym will be obtained by adding each of the subscale scores, with higher score indicating better health state.
Characterize patient characteristics initiating treatment with PI3K-inhibitors | 2 years
  Patient demographics, medical and disease history, prior therapies, and dosing regimen
Measure Time to Next Treatment (TTNT) | 2 years
  The length of time from the date the patient initiates PI3K-inhibitor treatment to the date of initiating the next line of therapy.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - CARTI Cancer Center, Little Rock, Arkansas
  - Joliet Oncology-Hematology Associates, LTD, Joliet, Illinois
  - Goshen General Hospital, Goshen, Indiana
  - McFarland Clinic,PC, Ames, Iowa
  - St. Agnes Hospital, Baltimore, Maryland
  - Regional Cancer Care Associates LLC, Bethesda, Maryland
  - Hattiesburg Clinic, PA, Hattiesburg, Mississippi
  - Capital Region Medical Center, Jefferson City, Missouri
  - Oncology Hematology Associates, Springfield, Missouri
  - NY Cancer and Blood Specialists, Port Jefferson Station, New York
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin